CLINICAL TRIAL: NCT07230938
Title: The Influence of Cervical Proprioception Deficits on Postural Stability in Patients With Cervical Spondylosis
Brief Title: Effects of Neck Proprioception Impairment on Balance in Cervical Spondylosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Aisha Mourad, principal investigator, MSc candidate, Delta University for Science and Technology
Other Study IDs: F.P.T250794
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Postural Stability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pedobarography system (foot pressure plateform) — Pedobarography system (foot pressure plateform) for Postural Stability assessment will be used to assess Postural stability. the pedobarographic analysis will be delivered using the FreeMed Professional platform (Sensor Medica, Rome, Italy). It evaluates the distribution of foot pressure on the ground.Three components make up the platform: a central mat with resistance sensors and two passive mats at either end that form a walking path. The platform is connected to a computer, to which all data is displayed and processed using FreeStep software
  Other Names: FREEMED baropodometric platform and FREESTEP software -v.2.01.054
Device: overhead laser pointer — laser pointer for Cervical proprioception device will be used to assess cervical proprioception by preforming Cervical joint position error (JPE) test

SUMMARY:
This observational cross-sectional study aims to investigate the impact of cervical proprioception deficits on postural stability in patients with cervical spondylosis. Using pedobarographic analysis, the study will assess static balance parameters in affected individuals. The main question it aims to answer is: Does Cervical proprioception deficits affect postural stability in patients with cervical spondylosis measured by pedobarographic parameters?

DETAILED DESCRIPTION:
This cross-sectional observational study intends to investigate the association between cervical proprioception and postural stability in people with cervical spondylosis. Cervical proprioception promotes posture regulation by providing sensory feedback to the central nervous system. Alterations in cervical joint position sensation caused by degenerative alterations can have a negative impact on balance.

Eighty participants with clinically diagnosed cervical spondylosis will be recruited. Each participant will undergo a single evaluation session that includes cervical joint position error testing and postural stability assessment using pedobarographic analysis. Data will be collected on center of pressure sway, weight distribution, and balance parameters under various conditions.

so this study findings can help physical therapists, rehabilitation experts, and clinicians design protocols to improve proprioceptive input and postural control in people with cervical spondylosis. Furthermore, early diagnosis of proprioceptive deficits by pedobarography may enable preventive actions and lower the incidence of falls and related morbidity in this population.

ELIGIBILITY:
Inclusion Criteria:

* Eighty-two patients with cervical spondylosis, the patient will be diagnosed and referred by physician.
* Mild to moderate cervical disability according to neck disability index( MacDermid et al., 2009).
* Age ranges from 25 to 45 years.
* Body mass index from 18.5 - 24.9.

Exclusion Criteria:

* The patients will be excluded if they have one of the following:
* visual or vestibular sensory disorders or cerebellar disease.
* Cervical myelopathy.
* Patients with previous cervical surgery.
* inflammatory diseases involving cervical spine such as rheumatoid arthritis or ankylosing spondylitis.
* History of cervical trauma including whiplash associated disorders (WAD).
* History of cervical tumors.
* History of ankle instability.
* No previous foot and ankle surgery.

Ages: 25 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Eighty-two patients with cervical spondylosis will represent the sample of this study. They will be selected from the outpatient clinic of Faculty of Physical Therapy, Delta University. All the patients will sign a consent form before starting the study
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Postural stability measured using a foot pressure platform | Single assessment at baseline (Day 1)
  Postural stability will be assessed by measuring postural sway using a force platform (stabilometer) under two conditions (eyes open and eyes closed). The primary variable will be the ellipse surface area (mm²) representing the center of pressure sway.

SECONDARY OUTCOMES:
Cervical joint position error (JPE) measured using overhead laser pointer | Single assessment at baseline (Day 1)
  Cervical proprioception will be measured using a laser pointer repositioning test. Participants will perform active neck movements and attempt to return to the neutral position with eyes closed. The average deviation (in degrees) from the starting point over three trials will be recorded. Errors greater than 4.5° will indicate proprioceptive impairment